CLINICAL TRIAL: NCT06229990
Title: Protocol Based-furosemide Stress Test Versus Standard Care to Evaluate Renal Recovery During Continuous Renal Replacement Therapy: A Randomized Controlled Trial
Brief Title: Protocol Based-furosemide Stress Test Versus Standard Care to Evaluate Renal Recovery During Continuous Renal Replacement Therapy
Acronym: PAUSE-CRRT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Prit Kusirisin, MD, Principal investigator, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MED-2566-0034
Record Dates: First submitted 2024-01-01; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Acute Kidney Injury
Keywords: Acute kidney injury; Continuous renal replacement therapy; Furosemide stress test; Critical care; CRRT
MeSH Terms: conditions — Acute Kidney Injury | interventions — Furosemide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protocol based-furosemide stress test (Experimental): Furosemide at 1.5 mg/kg intravenously
  Interventions: Drug: Furosemide Injection
- Standard care (No Intervention): Standard CRRT care without furosemide use during treatment.

INTERVENTIONS:
Drug: Furosemide Injection — After taking furosemide at 1.5 mg/kg intravenously, if the urine output exceeds 200 mL within 2 hours, the patients are going to withhold CRRT. But if there is no response, the titration of furosemide to 2.5 mg/kg and 3.5 mg/kg every 6 hours is scheduled according to the urine output >200 mL in 2 hours (not exceeding 250 mg).
  Other Names: Furosemide stress test
  Arms: Protocol based-furosemide stress test

SUMMARY:
Currently, continuous renal replacement therapy (CRRT) is the main modality for renal support in critically ill patients with hemodynamic instability. Most studies have investigated the timing of RRT initiation. However, prolonged CRRT demonstrated the association of many unexpected events, such as catheter-related complications, catheter-related blood stream infection, hypotension, hypothermia, tachycardia, and atrial fibrillation. Up to now, there is a lack of evidence regarding the timing of withholding CRRT. The furosemide stress test (FST) is a tool that is easy to use and has more availability. The investigators aimed to apply FST to evaluate renal recovery compared with standard treatment in critically ill patients undergoing CRRT.

ELIGIBILITY:
Inclusion Criteria:

* Adult 20 year of age or older
* Acute kidney injury (AKI) stage 3 according to Kidney Disease Improving Global Outcomes (KDIGO) classification with oliguria (urine <400 ml/day)
* Initiate CRRT in ICU (medical ICU, surgical ICU, cardiac care unit) for at least 48 hours (time for initiation and modality of CRRT can adjust by clinician)

Exclusion Criteria:

* Use any inotropic drug (norepinephrine, epinephrine, dopamine, dobutamine)
* Blood urea nitrogen (BUN) >80 mg/dL
* Serum K <3.5 or >5 mmol/L
* Arterial potential of Hydrogen (pH) <7.3
* Serum bicarbonate (HCO3) <15 mmol/L
* Urine volume <400 or >2,100 mL/day
* Urine creatinine clearance (CrCl) at 6 hours >20 mL/min
* Previous chronic kidney disease (CKD) stage 5 or estimated glomerular filtration rate (eGFR) <15 mL/min/1.73 m2
* Previous RRT within 14 days
* Kidney transplantation
* Obstructive etiology for AKI
* Toxin/drug that necessitates RRT
* Allergy to furosemide
* Moribund with expected death within 24 hours
* Pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-07 (Estimated); Study Completion 2024-06-07 (Estimated)

PRIMARY OUTCOMES:
% of patients with Renal recovery | 5 days
  Free of RRT for at least 5 days

SECONDARY OUTCOMES:
% of patients with Mortality | 28 days
  28 days all cause mortality and in-hospital mortality
RRT free days | 28 days
  No need to restart RRT
Day of Hospitalization | 28 days
  Length of hospital stay and ICU stay
Ventilator-free day | 28 days
  Number of mechanical ventilator-free day
% of complication | 28 days
  CRBSI, electrolyte imbalance, urine output
Cost of RRT during hospitalization | 28 days
  The cost of RRT since the initiation until the end of RRT during hospitalization in US dollar and Thai Baht unit

CONTACTS AND LOCATIONS:
Locations (1):
- Chiang Mai University, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Park S, Lee S, Jo HA, Han K, Kim Y, An JN, Joo KW, Lim CS, Kim YS, Kim H, Kim DK. Epidemiology of continuous renal replacement therapy in Korea: Results from the National Health Insurance Service claims database from 2005 to 2016. Kidney Res Clin Pract. 2018 Jun;37(2):119-129. doi: 10.23876/j.krcp.2018.37.2.119. Epub 2018 Jun 30. PMID 29971207
- [Result] Gaudry S, Hajage D, Schortgen F, Martin-Lefevre L, Pons B, Boulet E, Boyer A, Chevrel G, Lerolle N, Carpentier D, de Prost N, Lautrette A, Bretagnol A, Mayaux J, Nseir S, Megarbane B, Thirion M, Forel JM, Maizel J, Yonis H, Markowicz P, Thiery G, Tubach F, Ricard JD, Dreyfuss D; AKIKI Study Group. Initiation Strategies for Renal-Replacement Therapy in the Intensive Care Unit. N Engl J Med. 2016 Jul 14;375(2):122-33. doi: 10.1056/NEJMoa1603017. Epub 2016 May 15. PMID 27181456
- [Result] Zarbock A, Kellum JA, Schmidt C, Van Aken H, Wempe C, Pavenstadt H, Boanta A, Gerss J, Meersch M. Effect of Early vs Delayed Initiation of Renal Replacement Therapy on Mortality in Critically Ill Patients With Acute Kidney Injury: The ELAIN Randomized Clinical Trial. JAMA. 2016 May 24-31;315(20):2190-9. doi: 10.1001/jama.2016.5828. PMID 27209269
- [Result] Barbar SD, Clere-Jehl R, Bourredjem A, Hernu R, Montini F, Bruyere R, Lebert C, Bohe J, Badie J, Eraldi JP, Rigaud JP, Levy B, Siami S, Louis G, Bouadma L, Constantin JM, Mercier E, Klouche K, du Cheyron D, Piton G, Annane D, Jaber S, van der Linden T, Blasco G, Mira JP, Schwebel C, Chimot L, Guiot P, Nay MA, Meziani F, Helms J, Roger C, Louart B, Trusson R, Dargent A, Binquet C, Quenot JP; IDEAL-ICU Trial Investigators and the CRICS TRIGGERSEP Network. Timing of Renal-Replacement Therapy in Patients with Acute Kidney Injury and Sepsis. N Engl J Med. 2018 Oct 11;379(15):1431-1442. doi: 10.1056/NEJMoa1803213. PMID 30304656
- [Result] STARRT-AKI Investigators; Canadian Critical Care Trials Group; Australian and New Zealand Intensive Care Society Clinical Trials Group; United Kingdom Critical Care Research Group; Canadian Nephrology Trials Network; Irish Critical Care Trials Group; Bagshaw SM, Wald R, Adhikari NKJ, Bellomo R, da Costa BR, Dreyfuss D, Du B, Gallagher MP, Gaudry S, Hoste EA, Lamontagne F, Joannidis M, Landoni G, Liu KD, McAuley DF, McGuinness SP, Neyra JA, Nichol AD, Ostermann M, Palevsky PM, Pettila V, Quenot JP, Qiu H, Rochwerg B, Schneider AG, Smith OM, Thome F, Thorpe KE, Vaara S, Weir M, Wang AY, Young P, Zarbock A. Timing of Initiation of Renal-Replacement Therapy in Acute Kidney Injury. N Engl J Med. 2020 Jul 16;383(3):240-251. doi: 10.1056/NEJMoa2000741. PMID 32668114
- [Result] Gaudry S, Hajage D, Martin-Lefevre L, Lebbah S, Louis G, Moschietto S, Titeca-Beauport D, Combe B, Pons B, de Prost N, Besset S, Combes A, Robine A, Beuzelin M, Badie J, Chevrel G, Bohe J, Coupez E, Chudeau N, Barbar S, Vinsonneau C, Forel JM, Thevenin D, Boulet E, Lakhal K, Aissaoui N, Grange S, Leone M, Lacave G, Nseir S, Poirson F, Mayaux J, Asehnoune K, Geri G, Klouche K, Thiery G, Argaud L, Rozec B, Cadoz C, Andreu P, Reignier J, Ricard JD, Quenot JP, Dreyfuss D. Comparison of two delayed strategies for renal replacement therapy initiation for severe acute kidney injury (AKIKI 2): a multicentre, open-label, randomised, controlled trial. Lancet. 2021 Apr 3;397(10281):1293-1300. doi: 10.1016/S0140-6736(21)00350-0. PMID 33812488
- [Result] Akhoundi A, Singh B, Vela M, Chaudhary S, Monaghan M, Wilson GA, Dillon JJ, Cartin-Ceba R, Lieske JC, Gajic O, Kashani K. Incidence of Adverse Events during Continuous Renal Replacement Therapy. Blood Purif. 2015;39(4):333-9. doi: 10.1159/000380903. Epub 2015 May 22. PMID 26022612
- [Result] Chawla LS, Davison DL, Brasha-Mitchell E, Koyner JL, Arthur JM, Shaw AD, Tumlin JA, Trevino SA, Kimmel PL, Seneff MG. Development and standardization of a furosemide stress test to predict the severity of acute kidney injury. Crit Care. 2013 Sep 20;17(5):R207. doi: 10.1186/cc13015. PMID 24053972
- [Result] Lumlertgul N, Peerapornratana S, Trakarnvanich T, Pongsittisak W, Surasit K, Chuasuwan A, Tankee P, Tiranathanagul K, Praditpornsilpa K, Tungsanga K, Eiam-Ong S, Kellum JA, Srisawat N; FST Study Group. Early versus standard initiation of renal replacement therapy in furosemide stress test non-responsive acute kidney injury patients (the FST trial). Crit Care. 2018 Apr 19;22(1):101. doi: 10.1186/s13054-018-2021-1. PMID 29673370
- [Result] Lewis M, Bromley K, Sutton CJ, McCray G, Myers HL, Lancaster GA. Determining sample size for progression criteria for pragmatic pilot RCTs: the hypothesis test strikes back! Pilot Feasibility Stud. 2021 Feb 3;7(1):40. doi: 10.1186/s40814-021-00770-x. PMID 33536076